CLINICAL TRIAL: NCT00423995
Title: Study of the Decongestant Effect of the Combination of Loratadine and Montelukast Compared With Placebo in SAR Subjects Exposed to Pollen in an Environmental Exposure Unit
Brief Title: Effect of Loratadine/Montelukast Combination on Congestion in SAR Patients Exposed to Pollen in an EEU (Study P04822)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04822
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Loratadine/montelukast combination

SUMMARY:
This is study of LMC, phenylephrine, and placebo in subjects with SAR. There are three visits: At Visit 1, subjects will be evaluated for participation and, if they qualify, will attend Visit 2 for priming. At Visit 2, ragweed pollen will be fed continuously and dispensed into the environmental exposure unit to induce an allergic reaction. Pollen counts will be monitored and recorded. During the priming visit(s), subjects will be evaluated to determine if they qualify. If qualified, they will return for Visit 3, where ragweed pollen will be fed continuously and dispensed into the environmental exposure unit to induce an allergic reaction. Pollen counts will be monitored and recorded as in the Priming Session. Subjects will complete symptom evaluations and if qualified, they will receive study medication and remain in the environmental exposure unit where symptoms will be evaluated for 8 hours after dosing. PNIF will be evaluated only during the treatment session. Four nasal symptoms (rhinorrhea, nasal congestion, sneezing, and nasal itching) and three non-nasal symptoms (itching/burning eyes, tearing/watery eyes, and itching of ears/palate) will be evaluated. Adverse events will be collected throughout the study to assess safety and tolerability, and vital signs will be collected at Visit 1 and at the end of Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 years or greater, of either sex, any race.
* A history of SAR due to ragweed for at least two consecutive ragweed seasons, as diagnosed by the investigator, another physician, or subject-provided history.
* Positive skin prick test to ragweed allergen to be used in the EEU, unless previously done within 12 months
* Minimum scores (diary evaluation time) must be achieved during pollen exposure during both a Priming Visit and the Treatment Visit:
* A negative urine pregnancy test at Screening and prior to randomization at the Treatment Visit for all female subjects of childbearing potential.
* Use of a medically accepted method of birth control.
* In the judgment of the investigator, good health and freedom from any clinically significant disease (other than SAR) that would interfere with the study schedule or procedures, or compromise the subject's safety.
* The appropriate washout times from the prohibited medications.

Exclusion Criteria:

* Pregnancy, intention of becoming pregnant, or lactation.
* A situation or any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Use of any investigational drugs, including placebo, within 30 days of Screening and for the duration of the study.
* Current participation in any other clinical study.
* Staff personnel directly involved with this study.
* Dependence (in the opinion of the investigator) upon nasal, oral, or ocular decongestants, nasal topical antihistamines, or nasal steroids.
* Nasal structural abnormalities, including large nasal polyps or marked septal deviation, that cause greater than 50% obstruction of nasal airflow.
* Previous enrollment (ie, signed informed consent) into this study.
* History of rhinitis medicamentosa.
* A history of anaphylaxis or severe or serious reaction to skin testing.
* A known potential for hypersensitivity, allergy, or idiosyncratic reaction to the study drugs or excipients.
* Narrow-angle glaucoma, increased intraocular pressure, urinary retention, hypertension, severe coronary artery disease, ischemic heart disease, diabetes mellitus, hyperthyroidism, renal impairment, or prostatic hypertrophy; current treatment with monoamine oxidase (MAO) inhibitors.
* An upper or lower respiratory tract infection within 28 days (4 weeks) before Priming (Visit 2) and thereafter.).
* History of a positive test for HIV, TB (not due to vaccination), and hepatitis B (not due to vaccination) or C.
* Asthma that requires medication other than occasional (<= 3 uses per week) use of an inhaled short-acting beta-2 agonist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2007-03-01 (Actual); Study Completion 2007-03-10 (Actual)

REFERENCES:
- [Result] Day JH, Briscoe MP, Ratz JD, Danzig M, Yao R. Efficacy of loratadine-montelukast on nasal congestion in patients with seasonal allergic rhinitis in an environmental exposure unit. Ann Allergy Asthma Immunol. 2009 Apr;102(4):328-38. doi: 10.1016/S1081-1206(10)60339-0. PMID 19441605